CLINICAL TRIAL: NCT03450304
Title: Lung Perfusion Measured With Dual-Energy CT (DECT) in Patients With Chronic Thromboembolic Pulmonary Hypertension (CTEPH): Comparative Study With Right Heart Catheterization and Ventilation/Perfusion Scintigraphy (V/Q)
Brief Title: Lung Perfusion Measured With Dual-Energy CT in Patients With Chronic Thromboembolic Pulmonary Hypertension: Comparative Study With Right Heart Catheterization and V/Q
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Sergio Criales Vera (Unknown); Mariana Díaz Zamudio (Unknown); Nayeli Zayas Hernández (Unknown); Eric Kimura Hayama (Unknown); Regina De La Mora (Unknown); Tomás Pulido Zamudio (Unknown)
Responsible Party: Principal Investigator, César Cristancho rojas, Resident, Instituto Nacional de Cardiologia Ignacio Chavez
Other Study IDs: PT-17-050
Record Dates: First submitted 2018-02-22; First posted 2018-03-01 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Multidetector Computed Tomography; Pulmonary Embolism and Thrombosis; Hypertension Pulmonary Secondary
Keywords: Multidetector Computed Tomography; Pulmonary Embolism; Hypertension Pulmonary Secondary
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A comparative, observational, cross-sectional and prolective diagnostic test study, including patients that have had a right heart catheterization and were referred for a CT pulmonary angiography as part of their imaging workup protocol for pulmonary hypertension.

Dual-energy computed tomography (DECT) pulmonary angiography was performed on each patient to obtain perfusion maps and do a quantitative analysis. Segments with and without perfusion defects according to significant differences in the quantitative values, were defined as compatible or not with chronic thromboembolism.

To assess the accuracy of the method and evaluate its performance, these results were compared with the sole results from the right heart catheterization, known to be the gold standard diagnostic tool.

DETAILED DESCRIPTION:
a comparative, observational, cross-sectional and prolective diagnostic test study is conducted, including consecutive patients from the pulmonary hypertension clinic at our institution, from March 2017 to October 2018. Patients that have had a right heart catheterization and were referred for a CT pulmonary angiography as part of their imaging workup protocol. (The minimum sample size calculated is 26 patients).

DECT pulmonary angiography (256-slice and double-source CT scanner) was performed on each patient. Obtaining perfusion maps and doing a quantitative analysis by circular regions of interest (ROI) and iodine-related attenuation values (IRA) on each lung segment. Then, according to the finding in right heart catheterization, a comparison will be made between to groups: segments with and without perfusion defects, in order to find significant differences in the quantitative.

To assess the accuracy of the method and evaluate its performance, these results were later compared with the sole results from the right heart catheterization.

ROC curves were plotted to extract possible decision thresholds of the IRA values to classify perfusion as normal or deficient with this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the pulmonary hypertension clinic at our institution who have had right heart catheterization and were referred for a pulmonary CT angiography as part of their imaging workup protocol.

Exclusion Criteria:

* creatinine > 1.5 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients from the pulmonary hypertension clinic at our institution, from July 2017 to October 2018
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Lung perfusion measured with Dual-Energy CT (DECT) in patients with Chronic Thromboembolic Pulmonary Hypertension (CTEPH) | cross-sectional (one measurement). The minimum sample size calculated is 26 patients, which with the amount of patients handled in the pulmonary hypertension clinic at our institution is expect to reach in 16 months or before through study completion
  The objective is to evaluate lung perfusion quantification by DECT in patients with Chronic Thromboembolic Pulmonary Hypertension and compare findings with digital subtraction angiography with right heart catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiología Dr. Ignacio Chávez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
by request by mail